CLINICAL TRIAL: NCT04209946
Title: A Multicenter, Randomized Trial of Preterm Infants Receiving Caffeine and Less Invasive Surfactant Administration Compared to Caffeine and Early Continuous Positive Airway Pressure (CaLI Trial)
Brief Title: Early Caffeine and LISA Compared to Caffeine and CPAP in Preterm Infants
Acronym: CaLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other); Loma Linda University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CaLI
Record Dates: First submitted 2019-12-13; First posted 2019-12-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-03

CONDITIONS: Premature Lungs; Respiratory Distress Syndrome; Surfactant Deficiency Syndrome Neonatal
Keywords: Premature Infants; Respiratory Distress Syndrome; Less Invasive Surfactant administration; Continuous Positive Airway Pressure (CPAP)
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis; Premature Birth | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Less Invasive Surfactant Administration (LISA) (Active Comparator): Infants that are spontaneously breathing with a normal heart rate will be randomized to receive prophylactic surfactant (Curosurf 2.5 mL/kg, based on estimated fetal weight) by the LISA procedure in the first 2 hours of life, using a conventional or video laryngoscope and a small flexible 16 gauge angiocatheter. Any repeat dosing for surfactant will be based on clinical indication at the physician discretion by the conventional endotracheal approach.
  Interventions: Procedure: Less Invasive Surfactant Administration LISA
- Continuous Positive Airway Pressure (CPAP) (Active Comparator): Infants that are spontaneously breathing with a normal heart rate will be randomized to early Continuous Positive Airway Pressure (CPAP).
  Interventions: Procedure: Continuous Positive Airway Pressure CPAP

INTERVENTIONS:
Procedure: Less Invasive Surfactant Administration LISA — Laryngoscopy with insertion of a small 16 gauge angiocatheter to administer FDA approved Surfactant, during spontaneous respirations.
  Arms: Less Invasive Surfactant Administration (LISA)
Procedure: Continuous Positive Airway Pressure CPAP — Infant will remain on CPAP Therapy during spontaneous respirations
  Arms: Continuous Positive Airway Pressure (CPAP)

SUMMARY:
This study is being conducted to determine whether prophylactic administration of surfactant by the Less Invasive Surfactant Administration (LISA) method reduces the need for mechanical ventilation in the first 72 hours of life when compared to early Continuous Positive Airway Pressure (CPAP) alone.

DETAILED DESCRIPTION:
In order to allow for initial stabilization on CPAP, infants will be randomized by 1 hour of life. Consented infants that are assessed by a provider as clinically stable (i.e. HR> 100 bpm) and spontaneously breathing on CPAP will be randomized by computer generated randomization cards placed in opaque envelopes.

Randomization will be stratified by gestational age (24-26+6 weeks and 27-29+6 weeks) and labeled as such on each envelope. Multiples will be randomized to the same treatment group for ease of consent and family considerations.

Infants randomized to LISA will receive surfactant (Curosurf 2.5 mL/kg, based on estimated fetal weight) and must be given in the first 2 hours of life using a conventional or video laryngoscope and a small flexible 16 gauge angiocatheter.

All sites have agreed on using senior level physicians or practitioners that have prior experience with the LISA method. An orogastric tube will be placed into the stomach prior to laryngoscopy and the contents aspirated after the procedure to document any esophageal surfactant administration.

Infants randomized to early CPAP will be managed according to unit practice for preterm infants on CPAP.

Caffeine Administration:

If randomized to LISA, caffeine will be given prior to the LISA procedure. In contrast, if randomized to CPAP, caffeine will be given soon after birth. If infants in the CPAP group meet intubation criteria, and the loading dose of caffeine has not been administered, to avoid delay in intubation, caffeine will be given no later than thirty minutes after intubation.

As an unblinded trial it is critical that both groups are standardized to avoid bias towards one arm for intubation/treatment failure. Therefore, strict delivery room/NICU criteria will be used.

In the Delivery Room, criteria for intubation will be as specified in the Neonatal Resuscitation Program guidelines (7th Ed) and will include:

1. Chest compressions
2. Ineffective respiration
3. Prolonged positive pressure ventilation (PPV)
4. Prolonged hypoxia

In the Neonatal Intensive Care Unit (NICU), randomized infants in both groups will only be intubated if they meet strict failure criteria :

1. CPAP level of 6-8 cmH2O and FiO2> 0.40 required to maintain oxygen saturation >90% for 2 hours after randomization
2. pH of 7.15 or less OR a partial pCO2 >65 mmHg on any (2) blood gas (arterial/capillary/ or venous) at least 2 hours after randomization in the first 72 hours of life.
3. Continued Apnea/Bradycardia/Desaturation events despite nasal intermittent minute ventilation (NIMV) mode of ventilation.

Infants intubated prior to randomization will be excluded. Infants not consented prior to birth will also be excluded to avoid bias in patient selection.

For pragmatic purposes sites will be able to use their standard approach for non-invasive ventilation (NCPAP or NIMV).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born at 24 to 29+6 weeks gestation
* Informed consent obtained (antenatal)
* Infant is spontaneously breathing on CPAP of 5-8 cmH2O and maintaining a normal heart rate (HR>100 Bpm)

Exclusion Criteria:

* Declined consent
* Infants with known congenital anomalies
* Unstable immediately after birth, requiring intubation in the delivery room

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects requiring endotracheal intubation between the two groups (LISA vs CPAP) in the first 72 hours of life | Within 72 hours of life
  Required intubation or meeting respiratory failure criteria of having a pCO2 greater than 65 mm Hg or an FiO2 greater than 0.4 for more than 2 hours in the first 72 hours of life

SECONDARY OUTCOMES:
Duration of mechanical ventilation and/or CPAP | Through study completion at discharge, up to 6 months of corrected gestational age
  Number of days on mechanical ventilation and/or CPAP
Oxygen at 36 weeks corrected age | Up to 40 weeks of corrected gestational age
  Requiring oxygen therapy greater than 0.21 at 36 weeks corrected age
Frequency of Grade III and IV intraventricular hemorrhage | Through study completion at discharge, up to 6 months of corrected gestational age
  Intraventricular hemorrhage (grades 3-4)
Neurodevelopment outcome at 24 months of corrected gestational age | Up to 2 years of corrected gestational age
  Neurodevelopmental assessments using the Bayley Scales of Infant Development 4th ed. will be done at 2 years of corrected corrected age (22-26 months) for subjects who were randomized at birth to receive surfactant by the LISA method versus CPAP alone.
Neurodevelopment outcome at 2 Years of Age | 22-26 months corrected gestational age
  Overall and Domain Scores- Ages and Stages, 3rd ed. Questionnaire
Need for repeat surfactant dosing | Up to 40 weeks of corrected gestational age
  Requiring more than one dose of surfactant

OTHER OUTCOMES:
Laryngoscopy attempt with the LISA procedure | Number of laryngoscopy attempts per Surfactant dose, up to 36 weeks of corrected gestational age
  Total number of laryngoscopy attempts to administer surfactant via the LISA procedure
Laryngoscopy attempt with endotracheal intubation | Number of laryngoscopy attempts per Surfactant dose, up to 36 weeks of corrected gestational age
  Total number of laryngoscopy attempts to administer surfactant via endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Loma Linda Medical Center, Loma Linda, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, particularly data that underlie the results reported in this article after deidentification will be available with other researchers, including data dictionaries for meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 36 months following article publication
Access Criteria: Data and publication are available at http://clinicaltrials.gov
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Gopel W, Kribs A, Ziegler A, Laux R, Hoehn T, Wieg C, Siegel J, Avenarius S, von der Wense A, Vochem M, Groneck P, Weller U, Moller J, Hartel C, Haller S, Roth B, Herting E; German Neonatal Network. Avoidance of mechanical ventilation by surfactant treatment of spontaneously breathing preterm infants (AMV): an open-label, randomised, controlled trial. Lancet. 2011 Nov 5;378(9803):1627-34. doi: 10.1016/S0140-6736(11)60986-0. Epub 2011 Sep 29. PMID 21963186
- [Background] Kribs A, Hartel C, Kattner E, Vochem M, Kuster H, Moller J, Muller D, Segerer H, Wieg C, Gebauer C, Nikischin W, Wense Av, Herting E, Roth B, Gopel W. Surfactant without intubation in preterm infants with respiratory distress: first multi-center data. Klin Padiatr. 2010 Jan-Feb;222(1):13-7. doi: 10.1055/s-0029-1241867. Epub 2010 Jan 18. PMID 20084586
- [Background] Isayama T, Iwami H, McDonald S, Beyene J. Association of Noninvasive Ventilation Strategies With Mortality and Bronchopulmonary Dysplasia Among Preterm Infants: A Systematic Review and Meta-analysis. JAMA. 2016 Aug 9;316(6):611-24. doi: 10.1001/jama.2016.10708. PMID 27532916
- [Background] Bhayat S, Kaur A, Premadeva I, Reynolds P, Gowda H. Survey of less Invasive Surfactant Administration in England, slow adoption and variable practice. Acta Paediatr. 2020 Mar;109(3):505-510. doi: 10.1111/apa.14995. Epub 2019 Sep 16. PMID 31471992
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Katheria AC, Leone TA. Changes in hemodynamics after rescue surfactant administration. J Perinatol. 2013 Jul;33(7):525-8. doi: 10.1038/jp.2012.166. Epub 2013 Jan 17. PMID 23328925
- [Background] Dekker J, Hooper SB, van Vonderen JJ, Witlox RSGM, Lopriore E, Te Pas AB. Caffeine to improve breathing effort of preterm infants at birth: a randomized controlled trial. Pediatr Res. 2017 Aug;82(2):290-296. doi: 10.1038/pr.2017.45. Epub 2017 May 17. PMID 28288150
- [Background] Kurepa D, Perveen S, Lipener Y, Kakkilaya V. The use of less invasive surfactant administration (LISA) in the United States with review of the literature. J Perinatol. 2019 Mar;39(3):426-432. doi: 10.1038/s41372-018-0302-9. Epub 2019 Jan 11. PMID 30635595
- [Derived] Katheria A, Ines F, Banerji A, Hopper A, Uy C, Chundu A, Coughlin K, Hutson S, Morales A, Sauberan J, Poeltler D, Dorner R, Rich W, Finer N. Caffeine and Less Invasive Surfactant Administration for Respiratory Distress Syndrome of the Newborn. NEJM Evid. 2023 Dec;2(12):EVIDoa2300183. doi: 10.1056/EVIDoa2300183. Epub 2023 Nov 21. PMID 38320499
- [Derived] Ines F, Hutson S, Coughlin K, Hopper A, Banerji A, Uy C, Finer N, Rich W, Morales A, Steen J, Katheria AC. Multicentre, randomised trial of preterm infants receiving caffeine and less invasive surfactant administration compared with caffeine and early continuous positive airway pressure (CaLI trial): study protocol. BMJ Open. 2021 Jan 22;11(1):e038343. doi: 10.1136/bmjopen-2020-038343. PMID 33483435